CLINICAL TRIAL: NCT02522962
Title: Innovative Physiotherapy and Coordination of Care for People With Multiple Sclerosis: a Randomised Controlled Trial and a Qualitative Study
Brief Title: Innovative Physiotherapy and Coordination of Care for People With MS: a RCT and a Qualitative Study
Acronym: GroupCoreSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Helse Nord (Industry); University of Tromso (Other); University Hospital of North Norway (Other); Hasselt University (Other); University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1715 REK
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
Keywords: physical therapy; group-based; core stability; balance; movement quality; somatosensory stimulation; coordination
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupCoreSIT (Experimental): Before the group training starts, the physiotherapist in charge of the group does a clinical assessment of each participant in order to individualise the training. Each training group will consist of three participants. The training sessions will last for 60 minutes, performed three days per week, for six weeks, between 10 am and 5 pm.
  Interventions: Behavioral: GroupCoreSIT
- Standard care (Active Comparator): The control group receive standard care, which means to follow their ordinary physiotherapy services and/or routines/activities. The content of standard care may vary, and will be recorded for all the participants.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: GroupCoreSIT — Each group session lasts for 60 minutes. The physiotherapist will chose from an "exercises bank" of 32 exercises, each having up 5 levels of difficulty that are described and illustrated by photos. All exercises demand core activation, emphasise normal movement and emphasise somatosensory integration, feed forward and feed back strategies essential for balance.10-12 repetitions for each exercise with good quality of movement will be performed. Every session will start with exploring standing balance and end with active stretching/active relaxation, re-exploring balance and instructions for home exercises. The participants will perform 30-minute of exercises, optional to divide into smaller intervals, at home two days per week when there are no organized group training.
  Other Names: Group based individualised stability training; Group based individualised balance training
  Arms: GroupCoreSIT
Behavioral: Standard care — The control group receive standard care, which means to follow their ordinary physiotherapy services and/or routines/activities. The content of standard care may vary, and will be recorded for all the participants.
  Arms: Standard care

SUMMARY:
This project comprises a two-arm randomized controlled trial (RCT) complemented by qualitative research on innovative group-based intervention for people with Multiple Sclerosis (MS) performed in the primary health care and organized in collaboration with the services provided by a hospital's outpatient clinic. The RCT will be conducted by Nordland Hospital Trust, Bodø (NLSH), in collaboration with UiT The Arctic University of Norway (UiT) and the Norwegian Centre for Integrated Care and Telemedicine, University Hospital North Norway (NST). The overall purpose of the RCT is to demonstrate whether high-intensity individualised group-based core stability training (GroupCoreSIT) performed by physiotherapists (PTs) in the primary health care has effect on balance, walking and activities of daily living (ADL) in people with MS compared to standard care. Changes in quality of life and costs will also be studied to conclude whether the intervention is cost-effective. The qualitative study contains three parts. The first part aims to investigate users' experiences from participating in the new group intervention and in standard care. The researchers will particularly focus on reflections regarding content, feasibility, potential changes in ADL, self-management, and continuity of care. The second part will investigate how the PTs act and interact with the group while conducting the intervention, particularly how individualization is carried out, and the PTs' reflections from participating in the education and performance of the intervention. The third part explores health professionals' reflections regarding coordination of care in people with MS.

DETAILED DESCRIPTION:
This research project first aims to compare the effects of high-intensity individualized group-based core stability training (GroupCoreSIT) for people with MS with standard care in the primary health care focusing on balance, walking, ADL, quality of life and cost-effectiveness. Secondly, the project aims to investigate patients' experiences from participating in the intervention and in standard care, particularly addressing reflections regarding content, relevance and feasibility, changes in ADL, continuity of care, self-management. The third aim is to investigate how the PTs act and interact with the group while conducting the intervention, particularly how individualization is carried out, and the PTs' reflections from participating in the education and performance of the intervention. Finally, changes in patients' pathways and coordination represent another main objective of this project.

The RCT: hypothesis, study outcomes and measures:

High-intensity individualised group-based core stability training performed at the municipal PTs' facilities, complemented by home exercises, will improve balance, walking, ADL, quality of life and cost-effectiveness. This is reflected in the primary and secondary outcomes.

RCT will be conducted in collaboration with the outpatient clinic for people with MS at the Nordland Hospital Trust, Bodø, together with six municipalities in Nordland County. The municipalities are included: Bodø, Rana, Meløy, Rødøy, Vågan and Fauske. The out-patient clinic agreed to recruit the participants by sending a written invitation to people with MS in the selected municipalities, fulfilling the inclusion criteria. Six PTs with expertise in neurological physiotherapy agreed to conduct the intervention. These PTs will attend a four days practical and theoretical training on the intervention, with 1-2 follow up videoconferences during the study.

A prospective RCT will be conducted, in which 72 persons with MS will participate, undergo a 6-week intervention, and be followed up for 6 months. Participants will be randomly assigned to two arms in a 1:1 ratio. Participants in the intervention arm A will be offered individualised group-based core stability training termed GroupCoreSIT at the PTs facilities, complemented with home exercises. Participants in the control arm B will be offered standard care. Significant improvements in outcomes are expected for the intervention arm compared to standard care. Randomisation will be stratified by European Disability Score Scale (EDSS) to minimize selection bias and preserve homogeneity between arms. Randomisation and data collation will be performed using Remote Data Entry (WebCRF), an Internet-based solution developed by the Norwegian University of Science and Technology (NTNU). The researchers aim to recruit all subjects within 5 months.

After enrolment, the PTs responsible for performing the intervention, will conduct an individual assessment of the participants in arm A as a basis for individualisation in the group based intervention.

Each training group will consist of three participants. The training sessions will last for 60 minutes, performed three days per week, for six weeks, between 10 am and 5 pm. A total of 32 exercises with up to 5 levels of difficulty are described and illustrated by photos, will be available in an "exercise bank". 10-12 repetitions for each exercise with good quality of movement will be performed. Every session will end with active stretching/active relaxation and instructions for home exercises. The participants will perform 30-minute of exercises, optional to divide into smaller intervals, at home two days per week when there are no organized group training.

Intervention arm A: the participants will perform the training program: GroupCoreSIT in the facilities of the municipal physiotherapist.

Control arm B: the participants in the control group will receive standard care, i.e. following their ordinary physiotherapy services and/or routines/activities.

Procedures and tests The trial will be restricted to patients who have volunteered and provided written informed consent in accordance with the Declaration of Helsinki and the Ethics Committee procedures.

At enrolment, a neurologist will do the EDSS screening, medical history, type of MS and medications. An appropriately trained PT, also blinded to the arm membership, will perform a standardized assessment for all the participants using relevant tests and provide the activity monitor. The following baseline information will be collected and then inserted electronically in the WebCRF system used also to randomize the patients:

1. Medical history, type of MS, EDSS, age, gender, weight, height, medications, physiotherapy during the previous 6 months.
2. Two primary outcomes measuring balance in sitting, standing and walking.
3. Nine secondary outcomes measuring balance, waling, activities of daily living (ADL), quality of life and physical activity At 1 week, 3 months and 6 months post intervention all the participants will undergo the same standardized assessment performed at baseline.

Exercise, activity and disease monitoring On a weekly basis all the participants will record: changes in medication, general wellbeing (qualitative self-score), exacerbations, and physical activities using a diary. The ActiGraph monitor will be used 1 week prior to intervention, 1 week post intervention and following the 3 and 6 months testing, demonstrated and delivered to the subjects by the test PT. In addition, participants in arm A will record: degree of exhaustion following group sessions (Borg scale) and home exercise completion (in the training diary).

An intention-to-treat analysis will be performed on all randomised subjects and will serve as the primary analysis for all outcomes in this study. The data analysis will be carried out using SPSS. Possible differences between the groups at baseline will be calculated by using independent sample t-test for continuous variables and chi-square for categorical variables. Primary outcomes, changes in balance and walking between the groups will be calculated by using independent sample t-test.

A cost-utility analysis will be conducted using healthcare system costs and quality adjusted life years (QALYs). QALYs will be calculated based on the answers of the Health Questionnaire (EQ-5D-3L) used to measure changes in patients' quality of life. The incremental cost-effectiveness ratio (ICER) will be computed as differential costs between intervention arm and standard arm over the study period, and differential QALYs. Healthcare utilisation (including hospitalisations, emergency department admissions, outpatients visits, examinations, primary care visits, rehabilitation) and related costs will be collected through the hospitals' electronic patient journal (DIPS), from the Norwegian Patient Registry and The Norwegian Health Economics Administration's (HELFO) system. This secondary outcome will provide relevant knowledge regarding new effective method in organising healthcare services. This can be used as a basis for decision making regarding large-scale implementation of rehabilitation.

Patients' experiences:

The patients' experiences with the intervention will be examined through qualitative research interviews. The interviews will be conducted on a sample of 8-10 participants from the intervention and the control arm twice; at the end of intervention and 6 months post intervention. In accordance with qualitative methods, the researchers will select the sample strategically to promote breadth and variety of data production. Variation in training groups, EDSS, age, gender and time since diagnosis are considered to be important. The interviews will take place in participants' homes or another convenient place in their municipality. The interview topics include: the first assessment/consultation, the group situation, content of training, intensity/quantity, pros and cons, home-exercises and ADL. The same number of subjects from the control group will be interviewed regarding their experiences with standard care, investigating the same topics. In order to provide insight into the users' experiences beyond the intervention period the scope for the second interviews is: retrospective reflections regarding wellbeing and coping with ADL in the period before, during and after the intervention, self-management, and continuity of care, pros and cons regarding the intervention and standard care. A theme-based interview guide will be used as well as audio recordings of the interviews. The material will be transcribed and analyzed using Systematic Text Condensation applying phenomenology of the body, enactive theory complemented by neurosciences as a theoretical framework.

Physiotherapists' performance of intervention and experiences:

What the PTs emphasize in their individual assessment prior to the first group session will be investigated through observation and videotaping of the assessment of one patient in each training group (12 observations). These observations will be complemented by qualitative research interview with the actual PT (12 interviews) to illuminate the PTs' reflections regarding the assessment, planning of the group sessions, choices of exercises and goals for the individual. To investigate how the PTs' tailor the intervention in situ, how they act and interact with the participants, one session in each group will be observed and videotaped (12 observations). To illuminate the PTs' reflections regarding education in the intervention, experiences from conducting it, particularly focusing on considerations regarding goal attainment, individualization in a group setting and home exercises, the PTs will be interviewed at the end of each training group period (12 interviews). An observation guide, a hand held video-camera and a theme-based interview guide will be used as well as audio recordings of the interviews. The material will be transcribed and analysed using Systematic Text Condensation applying phenomenology of the body, enactive theory complemented by neurosciences and practice knowledge as a theoretical framework.

Changes in patient's pathway and coordination of care:

In 2007 The Northern Norway Regional Health Authority (Helse Nord RHF) reported 650 persons with MS, the selected outpatient clinic has 300 persons enrolled, and prevalence and incidence in Nordland County have recently increased to a high risk area for MS. Courses for newly diagnosed persons have priority in the specialist care and current offer of complex rehabilitation, included high intensity physiotherapy is provided by the rehabilitation unit at UNN, The Rehabilitation Centre, the Kurbad of North Norway, Valnesfjord Rehabilitation Centre, supplemented by The National Hakadal MS centre. These institutions are currently characterised by long waiting lists. A system for early admission to neurological physiotherapy, and particularly to high intensity programs in the primary health care, is not established within the coordination of care for people with MS. Referral to municipality physiotherapy is not systematic, waiting lists in the primary health care are long, and services are often general and not specifically addressing the needs for people with MS.

To explore coordination of care between the outpatient clinics for people with MS and the municipalities regarding high intensity physiotherapy, qualitative interviews will be conducted with selected health personnel (MS-nurses, neurologists, PTs, a total of 8-10 subjects) at the hospitals' outpatient clinics and in municipalities (general practitioners, PTs, a total of 8-10 subjects), before the intervention (for the standard care) and after the RCT (for the new organizational model). The interviews will focus on structures for collaboration and content of service.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (McDonald's criteria)
* EDSS 1-6.5 (minimal symptoms - able to walk 20 minimum meter with two crutches)
* Minimum 14 days post exacerbation
* Age >18 years
* Capable to provide signed written informed consent

Exclusion Criteria:

* Pregnancy at enrolment
* Acute orthopedic conditions affecting balance and walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale modified Norwegian Version | Baseline
  The outcome measures sitting balance
Measure change in the outcome: Trunk Impairment Scale modified Norwegian Version | 1 week post intervention
  The outcome measures sitting balance
Measure change in the outcome: Trunk Impairment Scale modified Norwegian Version | 3 months post intervention
  The outcome measures sitting balance
Measure a change in the outcome: Trunk Impairment Scale modified Norwegian Version | 6 months post intervention
  The outcome measures sitting balance
Mini-Balance Evaluation Systems Test | baseline
  The outcome measures standing and walking balance
Measure a change in the outcome: Mini-Balance Evaluation Systems Test | 1 week post intervention
  The outcome measures standing and walking balance
Measure a change in the outcome:Mini-Balance Evaluation Systems Test | 3 months post intervention
  The outcome measures standing and walking balance
Measure a change in the outcome: Mini-Balance Evaluation Systems Test | 6 months post intervention
  The outcome measures standing and walking balance

SECONDARY OUTCOMES:
10-Meter Walk Test | Baseline
  The outcome measures the speed of 10 meter walking
Measure a change in the outcome: 10 Meter Walk Test | 1 week post intervention
  The outcome measures the speed of 10 meter walking
Measure a change in the outcome:10 Meter Walk Test | 3 months post intervention
  The outcome measures the speed of 10 meter walking
Measure a change in the outcome: 10 Meter Walk Test | 6 months post intervention
  The outcome measures the speed of 10 meter walking
2-Minutes Walk Test | Baseline
  The outcome measures the distance walked in 2 minutes
Measure a change in the outcome: 2-Minutes Walk Test | 1 week post intervention
  The outcome measures the distance walked in 2 minutes
Measure a change in the outcome:2-MinutesWalk Test | 3 months post intervention
  The outcome measures the distance walked in 2 minutes
Measure a change in the outcome:2-Minutes Walk Test | 6 months post intervention
  The outcome measures the distance walked in 2 minutes
Rivermead Visual Gait Assessment | Baseline
  The outcome measures quality of movement in walking
Measure a change in the outcome:Rivermead Visual Gait Assessment | 1 week post intervention
  The outcome measures quality of movement in walking
Measure a change in the outcome:Rivermead Visual Gait Assessment | 3 months post intervention
  The outcome measures quality of movement in walking
Measure a change in the outcome:Rivermead Visual Gait Assessment | 6 months post intervention
  The outcome measures quality of movement in walking
MS Walking Scale-12 | Baseline
  a self-report form with 12 questions where limitations in various aspects of walking in the past two weeks are detected.
Measure a change in the outcome:MS Walking Scale-12 | 1 week post intervention
  a self-report form with 12 questions where limitations in various aspects of walking in the past two weeks are detected.
Measure a change in the outcome:MS Walking Scale-12 | 3 months post intervention
  a self-report form with 12 questions where limitations in various aspects of walking in the past two weeks are detected.
Measure a change in the outcome: MS Walking Scale-12 | 6 months post intervention
  a self-report form with 12 questions where limitations in various aspects of walking in the past two weeks are detected.
Multiple Sclerosis Impact Scale-29 | Baseline
  A self-report form with 29 items which records limitations in various aspects of ADL
Measure a change in the outcome:Multiple Sclerosis Impact Scale-29 | 1 week post intervention
  A self-report form with 29 items which records limitations in various aspects of ADL
Measure a change in the outcome:Multiple Sclerosis Impact Scale-29 | 3 months post intervention
  A self-report form with 29 items which records limitations in various aspects of ADL
Measure a change in the outcome:Multiple Sclerosis Impact Scale-29 | 6 months post intervention
  A self-report form with 29 items which records limitations in various aspects of ADL
The Patient Global Impression of Change | 1 week post intervention
  a self-report form that measures the subject's perceptions of change
Measure a change in the outcome: Patient Global Impression of Change | 3 months post intervention
  a self-report form that measures the subject's perceptions of change
Measure a change in the outcome: Patient Global Impression of Change | 6 months post intervention
  a self-report form that measures the subject's perceptions of change
ActiGraph activity monitor. | baseline
  The outcome measures physical activity
Measure a change in the outcome:ActiGraph activity monitor. | 1 week post intervention
  The outcome measures physical activity
Measure a change in the outcome:ActiGraph activity monitor | 3 months post intervention
  The outcome measures physical activity
Measure a change in the outcome:ActiGraph activity monitor | 6 months post intervention
  The outcome measures physical activity
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Baseline
  The outcome measures the participants' health related quality of life.
Measure a change in the outcome:Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 1 week post intervention
  The outcome measures the participants' health related quality of life.
Measure a change in the outcome:Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 3 months post intervention
  The outcome measures the participants' health related quality of life.
Measure a change in the outcome:Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 6 months post intervention
  The outcome measures the participants' health related quality of life.
Health Questionnaire (EQ-5D-3L) | Baseline
  The outcome measures the participants' health quality of life.
Measure a change in the outcome:Health Questionnaire (EQ-5D-3L) | 1 week post intervention
  The outcome measures the participants' quality of life.
Measure a change in the outcome:Health Questionnaire (EQ-5D-3L) | 3 months post intervention
  The outcome measures the participants' quality of life.
Measure a change in the outcome:Health Questionnaire (EQ-5D-3L) | 6 months post intervention
  The outcome measures the participants' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Normann, PhD, Study Chair — Nordlandssykehuset HF
Locations (1):
- Physiotherapy department, Nordlandssykehuset HF, Bodø, Norway

REFERENCES:
- [Derived] Arntzen EC, Straume BK, Odeh F, Feys P, Zanaboni P, Normann B. Group-Based Individualized Comprehensive Core Stability Intervention Improves Balance in Persons With Multiple Sclerosis: A Randomized Controlled Trial. Phys Ther. 2019 Aug 1;99(8):1027-1038. doi: 10.1093/ptj/pzz017. PMID 30722036